CLINICAL TRIAL: NCT00118833
Title: Placebo-Controlled Trial of Hypericum Perforatum in the Treatment of Generalized Social Anxiety Disorder (GSAD)
Brief Title: St. John's Wort for the Treatment of Generalized Social Anxiety Disorder (GSAD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K23AT000583-01 (NIH)
Record Dates: First submitted 2005-07-07; First posted 2005-07-12 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Anxiety Disorders; Mental Health
Keywords: Social Anxiety Disorder; Social Phobia; Generalized Anxiety Disorder; Hypericum; St. John's wort; Medicine, Herbal; Complementary Therapies
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being; Phobia, Social; Generalized Anxiety Disorder | interventions — Hypericum extract LI 160

INTERVENTIONS:
Drug: Hypericum perforatum (St. John's wort)

SUMMARY:
This study will determine whether the herbal product St. John's wort is safe and effective in treating generalized social anxiety disorder (GSAD).

Study hypothesis: Hypericum perforatum (St. John's wort) is more effective in treating GSAD than placebo.

DETAILED DESCRIPTION:
The use of complementary and alternative medicine (CAM) has grown dramatically over the last decade. Botanical treatments originating from plants have become especially popular for treating conditions such as anxiety and depression. Evidence suggests that the botanical St. John's wort has neurochemical activity similar to that of conventional medications. However, research on the safety and effectiveness of St. John's wort is limited. This study will determine the safety and effectiveness of St. John's wort in treating GSAD, a serious condition characterized by intense fear of various social situations that may cause embarrassment.

Participants will be randomly assigned to receive either St. John's wort or placebo daily for 10 weeks. Self-report scales will be used to assess participants' GSAD symptoms at study entry and at study completion. Blood collection will occur at every weekly study visit to determine the levels of St. John's wort in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GSAD
* Brief Social Phobia Scale (BSPS) score of 20 or higher

Exclusion Criteria:

* Comorbid anxiety, depressive, or bipolar disorders
* Schizophrenia
* Cognitive impairment
* Substance abuse or dependence within 1 year prior to study entry
* Any unstable medical condition
* Clinically significant laboratory or electrocardiogram (EKG) abnormality
* Currently use psychotropic medications or may need psychotropic medication during the study
* Psychotherapy within 6 weeks prior to study entry
* Failed a previous trial of St. John's wort at doses of 1800 mg/day or greater
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2002-08; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression (CGI), designed to assess global severity of illness and change in the clinical condition over time

SECONDARY OUTCOMES:
Brief Social Phobia Scale (BSPS)
Liebowitz Social Anxiety Scale
Social Phobia Inventory (SPIN)
Self-Rating Depression Scale (SDS)
Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States